CLINICAL TRIAL: NCT01999829
Title: Prevention of Atrial Fibrillation Following Valvular Replacement With Cardiopulmonary Bypass: a Prospective, Randomized Clinical Study Comparing Oral Caffeine With Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-23; 2013-23 (Other: AP HM)
Record Dates: First submitted 2013-09-26; First posted 2013-12-03 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2015-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- citrate of caffeine (Experimental)
  Interventions: Drug: citrate of caffeine
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: citrate of caffeine
  Arms: citrate of caffeine
Drug: placebo
  Arms: placebo

SUMMARY:
Atrial fibrillation remains a major cause of morbidity following cardiac surgery with cardiopulmonary bypass. Many mechanisms have been implicated. Among then, adenosine, a strong endogenous vasodilating agent has been involved in cardiac surgery-induced atrial fibrillation, via A2A receptors modulation.

The effects of caffeine on the inducibility of atrial fibrillation are actually well-known, leading then to a significant reduction of atrial fibrillation. Moreover, a recent clinical study has demonstrated that coffee drinking was inversely associated with total and cause-specific mortality.

The investigators therefore examined the preventive effects of oral caffeine on valvular surgery with cardiopulmonary bypass-induced atrial fibrillation. The investigators also evaluated prospectively the influence of caffeine on adenosine plasma levels and A2A adenosine receptors modulation.

ELIGIBILITY:
Inclusion Criteria:

* Age = 18 years
* Surgery valvular settled(adjusted) (plasties or aortic replacement, mitral, tricuspid or mixed), under CEC
* Period of weaning in caffeine: limitation of the consumption of coffee(café), tea, chocolate, in a cup the day before the intervention
* Consent of the patients after information

Exclusion Criteria:

* Pregnant or breast-feeding women
* Women taking an oral contraception (half-life of the caffeine increased until 3 times)
* Minors(miners) or adults under guardianship
* Persons staying in a sanitary or social establishment
* Not profitable persons of a national insurance scheme
* Private persons of freedom
* Persons requiring a surgery of replacement valvular as a matter of urgency
* Patients having been treated(handled) by papaverine, dipyridamole, corticoids, immunosuppressors or antibiotics during six weeks preceding the date of inclusion
* Weighty patient lower than 50 kg or upper to 100 kg or having a body mass index upper to 29 Kg / m2
* Presence of an active infection, a chronic inflammatory pathology, a lung arterial high blood pressure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Decrease of 50 % of the incidence of atrial fibrillation | 24 MONTHS

SECONDARY OUTCOMES:
decrease in the use of anti-arrhythmic resuscitation | 24 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Lagier D, Nee L, Guieu R, Kerbaul F, Fenouillet E, Roux N, Giorgi R, Theron A, Grisoli D, Gariboldi V, Collart F, Bruder N, Velly L, Guidon C. Peri-operative oral caffeine does not prevent postoperative atrial fibrillation after heart valve surgery with cardiopulmonary bypass: A randomised controlled clinical trial. Eur J Anaesthesiol. 2018 Dec;35(12):911-918. doi: 10.1097/EJA.0000000000000824. PMID 29702502